CLINICAL TRIAL: NCT01646567
Title: A Double-Blind, Within-Subject Randomised, Placebo-Controlled, Proof of Concept, Comparison Study of SHP-141C Topical Cream in Psoriasis, Using the Microplaque Assay.
Brief Title: SHP-141C in Plaque Type Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TetraLogic Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHP-141C-002
Record Dates: First submitted 2012-07-11; First posted 2012-07-20 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Plaque Type Psoriasis
Keywords: psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Betamethasone Valerate; calcipotriene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- SHP-141C & Placebo & Calcipotriol & Betamethasone Valerate (Experimental): A 100 mg dose of SHP-141C cream at three concentrations (0.5%, 1.0% and 2.0%), a matched placebo cream and two reference treatments: Calcipotriol 0.005% cream and Betamethasone Valerate 0.02% cream, applied topically to a selected plaque on each subject, six times per week over 28 days for a total of 24 doses.
  Interventions: Drug: SHP-141C; Drug: Placebo to SHP-141C; Drug: Betamethasone Valerate; Drug: Calcipotriol

INTERVENTIONS:
Drug: SHP-141C — Topical Cream
  Other Names: SHAPE
Drug: Placebo to SHP-141C — Placebo Topical Cream
  Other Names: Placebo to SHAPE
Drug: Betamethasone Valerate — Topical cream, 0.02%
  Other Names: Celestone-M
Drug: Calcipotriol — Topical cream, 0.005%
  Other Names: Daivonex

SUMMARY:
The purpose of this study is to assess the safety, tolerability and clinical activity of the SHP-141C topical cream formulations in patients with plaque type psoriasis.

DETAILED DESCRIPTION:
Psoriasis is a chronic, relapsing immunoinflammatory disorder. Chronic plaque psoriasis is the most common (85% - 90%) type. Cutaneous features of individual plaques include circular with centrifugal expansion, induration with sharp demarcation from surrounding skin, erythema and hyperkeratosis. Psoriasis has a negative impact on physical and mental aspects of life that is similar to other major chronic conditions. The modalities of psoriasis treatments can be divided into four main categories: topical, phototherapy, systemic drug therapies and systemic biological treatments. The currently available treatments for psoriasis result in either disease suppression or disease remission.There are many treatment options for the management of psoriasis using topical modalities; however all are lacking with respect to patient satisfaction and durability of treatment. Most current topical treatments, and many treatments in development, are based on modifications of a steroid structure or on Vitamin D. Recent research has identified a broad role for histone deacetylase (HDAC) proteins in numerous signaling pathways critical to cancer cell survival, such as epigenetic inheritance, gene regulation, mitosis,signal transduction and importantly, inflammation. Theoretically modulation of HDAC could lead to clinical benefit in inflammatory diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Mild to moderate chronic plaque-type psoriasis.
2. psoriasis of at least one year.
3. Stable disease for at least two weeks prior to the commencement of study treatment.
4. One nominated target lesions must have areas of at least 86 x 57 mm2.
5. BMI of less than 35 kg/m2. -

Exclusion Criteria:

1. Dermatological Conditions

   * Subjects with erythrodermic, guttate, palmar, plantar or generalised pustular forms of psoriasis.
   * Subjects with scalp, palmar or plantar psoriasis only.
   * Subjects with any skin condition other than psoriasis, in particular eczema, cutaneous infections, significant sun damage or an inherited skin disorder (other than psoriasis).
2. Concurrent Medical Conditions

   * History of clinically significant intercurrent disease of any type (other than psoriasis).
   * A history of moderate or severe asthma during the last 10 years.
   * Major chronic inflammatory disease .
   * Congenital immunodeficiency or cancer prone syndrome.
   * History of abnormal bleeding tendencies or thrombophlebitis, or a history of Hepatitis B, Hepatitis C or HIV infection.
   * History of malignancy (other than adequately treated skin carcinoma or carcinoma-in-situ of the cervix).
3. Laboratory Status

   * Any evidence of organ dysfunction, which is confirmed on re-examination to be clinically significant (i.e. in the opinion of the Medical Officer would jeopardise the safety of the subject or impact on the validity of the study results),
   * A creatinine clearance of less than 75 mL/min.
   * Liver function test > 1.5 x upper limit of normal other than an isolated bilirubin.
   * Hepatitis B surface antigen, Hepatitis C antibody, HIV antibodies.
4. Treatment with any of the following within 4 weeks prior to the commencement of study treatment and for the duration of the study:

   * Systemic retinoids.
   * Immunosuppressant agents (e.g. methotrexate, cyclosporine, azathioprine, thioguanine prednisone, prednisolone, hydroxyurea or mycophenolate mofetil).
   * Phototherapy or photochemotherapy.
   * High potency topical corticosteroids.
   * "Alternative medicine" treatments for psoriasis.
   * Prolonged sun exposure or tanning bed use, which may in the opinion of the Investigator, modify disease activity.
5. Topical treatment of the 2 target lesions with any of the following within 2 weeks prior to commencement of study treatment and for the duration of the study

   * Moderate potency topical corticosteroids.
   * Vitamin D analogues and topical retinoids.
   * Keratolytics, coal tar and dithranol.
6. Concurrent Medications Subjects have received or anticipate receiving a new medicine (prescription, over-the-counter or herbal), given systemically or topically, within 14 days prior to the start of dosing. Subjects may be enrolled if stable on existing therapy (having been on it for at least 60 days) as determined by the Principal Investigator.
7. Hypersensitivity History of allergy and/or hypersensitivity to any of the stated ingredients of the formulations or other topical agents. A known hypersensitivity to lignocaine, or all surgical dressings that may be used in the study procedures.
8. Females who are lactating, pregnant or planning to become pregnant.
9. Drug and Alcohol Abuse History of, or current evidence of, abuse of alcohol or any drug substance, licit or illicit, or positive urine drug and alcohol screen for drugs of abuse and alcohol.
10. Psychiatric Disorder History of any psychiatric illness which may impair the ability to provide written informed consent
11. Participation in a research study within 30 days of the start of dosing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Local Plaque Severity Index (LPSI) | Baseline, day 15, day 33
  Measurement of plaque severity including erythema, induration, and desquamation.

SECONDARY OUTCOMES:
The number of patients with adverse events | daily to and including Day33
  Adverse event data for each subject will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Foley, Principal Investigator — The Alfred
Locations (1):
- Nucleus Network Limited, Melbourne, Victoria, Australia